CLINICAL TRIAL: NCT01700413
Title: Treatment of di Novo Acute Myeloid Leukemia With the Combination of Increasing Doses of Idarubicin, Cytarabine and Sensitization (Priming) With G-CSF. A Phase II Prospective Study of Toxicity and Efficacy.
Brief Title: Efficacy and Toxicity of Increasing Doses of Idarubicin, Cytarabine and G-CSF in Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other)
Collaborators: Ministry of Health, Spain (Other Government); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-CSF-2011-141
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Di Novo Acute Myeloid Leukemia
Keywords: acute; myeloid; leukemia; CETLAM; Idarubicin
MeSH Terms: conditions — Leukemia | interventions — Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Idarubicin (Experimental): Cohort 1: Idarubicin 14 mg/m2 (day 1-3), Cytarabine 200 mg/m2 (Days 1-7), G-CSF 150 mcg/m2/day Cohort 2: Idarubicin 16 mg/m2 (day 1-3), Cytarabine 200 mg/m2 (Days 1-7), G-CSF 150 mcg/m2/day Cohort 3: Idarubicin 18 mg/m2 (day 1-3), Cytarabine 200 mg/m2 (Days 1-7), G-CSF 150 mcg/m2/day
  Interventions: Drug: Idarubicin

INTERVENTIONS:
Drug: Idarubicin

SUMMARY:
While several studies have been reported with increasing doses of daunorubicin in the first line treatment of Acute Myeloid Leukemia (AML), there is no similar experience with idarubicin as initial treatment of AML.

As idarubicin is the most common treatment used for AML, it is needed to find the optimal dose for the combination of idarubicin, cytarabine and G_CSF, to explore if this combination improves the outcomes of current treatments for AML.

The aim of this dose-finding study is to find the optimal dose for the combination of idarubicin, cytarabine and G-CSF that could improve the response rate, reduce relapse and improve survival of patients with primary acute myeloid leukemia. This could be a significant advance in a field where treatment outcomes have stabilized in the last 15 years. This study will be the basis for further prospective, randomized, multicenter trial comparing idarubicin maximum tolerated dose, compared to standard treatment with idarubicin and cytarabine, including raising both arms in G-CSF. The dose of 12 mg/m2 will be administered as control arm in this future randomized study, which will investigate the benefit of enhanced dose identified as optimal in this phase II pilot study.

ELIGIBILITY:
Inclusion Criteria:

Informed consent signature Patients with newly diagnosed AML, classified according to WHO criteria. Age more than or equal to 18 and less than or equal to 70 years.

Exclusion Criteria:

Patients previously treated with chemotherapy for their AML other than hydroxyurea.

Acute promyelocytic leukemia with t (15; 17). Blast crisis of chronic myeloid leukemia. Leukemias that appear after other myeloproliferative neoplasms. Leukemias ensuing myelodysplastic syndromes after more than 6 months. Presence of other malignancies in activity. AML secondary to chemo-radiotherapy treatment for other malignancies. Abnormal renal and hepatic function, with creatinine value and / or bilirubin 2 times the normal limit value, except where the alterations are attributable to leukemia.

Patients with markedly reduced ejection fraction (less than 45%), symptomatic heart failure, or both of the normal value of the center.

Patients with serious concomitant psychiatric or neurological disease. HIV-positive. Pregnancy or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Rate of complete remissions (CR) | From 28 up to 56 days after first induction
  Identify the highest dose of idarubicin in combination with cytarabine and G-CSF that produces a CR rate equal to or greater than 65% with tolerable toxicity.

SECONDARY OUTCOMES:
Rate of patients with adverse events as a measure of safety and tolerability | Weekly during treatment, and on months 3 and 6 after complete response
  Hematologic toxicity Gastrointestinal and liver toxicity Cardiac Toxicity Fever and infection Pulmonary complications Duration of hospitalization Mortality and causes of death induction.
Duration of hospitalization | From the inclusion until 9 months after inclusion.
  Number of days in which the patient is hospitalized.
Mortality (as rate) related to study treatment | Weekly during treatment, 3 months after complete remission, 6 months after complete remission and 9 months after complete remission
  Causes of death, mortality related treatment, mortality in induction.
Relapse at 6 months | 6 months from complete remission, expected to be within 9 months from inclusion.
  Rate of patients that have relapsed within 6 months after complete remission.
Survival at 9 months from diagnosis | 9 months after diagnoses
  Rate of patients alive at 9 months after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Salut Brunet, MD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (5):
- Spain (5):
  - Hospital Universitari Germans Trias I Pujol de Badalona, Badalona, Badalona
  - Hospital de La Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospitals Vall D'Hebron, Barcelona, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia